CLINICAL TRIAL: NCT06584019
Title: The Effect of Range of Motion (ROM) Exercises Applied to Oncology Patients in the 6-12 Years Group on the Comfort Level and Vital Signs
Brief Title: The Effect of Range of Motion (ROM) exercıses on Comfort Level and vıtal sıgns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, aysel kokcudogan, Ph.D., Asst. Prof., Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-10840098-772.02-7434
Record Dates: First submitted 2024-07-19; First posted 2024-09-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Children With Cancer
Keywords: Range Of Motion exercises; cancer; pediatrics; comfort
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Range Of Motion applied group (Experimental): Children with cancer were given Range Of Motion exercises once a day for 5 days for approximately 20 minutes.
  Interventions: Other: Range Of Motion applied group
- Control group (No Intervention): Children with cancer in this group received no intervention.

INTERVENTIONS:
Other: Range Of Motion applied group — Range Of Motion was applied once a day for approximately 20 minutes for 5 days.
  Arms: Range Of Motion applied group

SUMMARY:
This experimental study aims to examine the effects of ROM (Range of Motion) exercises on comfort level and vital signs in children diagnosed with cancer.

DETAILED DESCRIPTION:
The sample of the study consisted of a total of 60 oncology patient children, 30 in the experimental group and 30 in the control group, between the ages of 6-12, who were hospitalized in the Pediatric Bone Marrow Transplant Unit and Pediatric Hematology Oncology Service of a state hospital. The data of the study were collected with the "Data Collection Form", "Life Findings Table" and "Comfort Scale in Children". Range of motion exercise applications continued once a day for 5 days a week for approximately 20 minutes. Fever, pulse, respiration, blood pressure, pain and comfort levels of the children were measured before and after the exercise. In the study, it was investigated whether Range of motion exercises have an effect on vital signs and comfort levels of children with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between 6 and 12 years of age.
* Patients diagnosed with oncology.
* Patients who agreed to participate in the study and whose consent was obtained from their parents.
* Patients who can communicate and are conscious.

Exclusion Criteria:

* Patients with fractures or orthopedic conditions that may limit exercise.
* Patients with serious cardiac problems that may prevent exercise.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Body temperature | For 5 days/ 2 times a day/ before and after a 20 minute range of motion.
  For 5 days, children's body temperature was taken 2 times before and after 20 minutes of Range Of Motion.
Pulse | For 5 days/ 2 times a day/ before and after a 20 minute range of motion.
  For 5 days, children's pulse was taken 2 times before and after 20 minutes of Range Of Motion.
Respiration | For 5 days/ 2 times a day/ before and after a 20 minute range of motion.
  For 5 days, children's Respiration was taken 2 times before and after 20 minutes of Range Of Motion.
Blood pressure | For 5 days/ 2 times a day/ before and after a 20 minute range of motion.
  For 5 days, children's systolic blood pressure and diastolic blood pressure was taken 2 times before and after 20 minutes of Range Of Motion.
Comfort | For 5 days/ 2 times a day/ before and after a 20 minute range of motion.
  For 5 days, children's comfort level was taken 2 times before and after 20 minutes of Range Of Motion.
  Pediatric Comfort Assessment Scale was used for measurement. It evaluates 5 parameters: sounds, motor movements, performance, facial expressions and other. Each item is evaluated on a 5-point Likert scale from 0 to 4 (0/Not Available, 1/No, 2/Somewhat, 3/Moderate, 4/Strong) from bad to good. Higher scores indicate a higher level of comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Aysel Kokcu Dogan, Asst. Prof., Study Director — Istanbul Medipol University faculty member
Locations (1):
- Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No